CLINICAL TRIAL: NCT01214161
Title: Intracervical Two Percent Lidocaine Gel as an Analgesic During Intrauterine Device Insertion: A Randomized Controlled Trial
Brief Title: Intracervical Lidocaine Gel for IUD Insertional Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Anne Davis, Associate Professor of Obstetrics and Gynecology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AAAE9330
Record Dates: First submitted 2010-09-29; First posted 2010-10-04 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: Pain
Keywords: IUD; Lidocaine gel
MeSH Terms: conditions — Pain | interventions — phenylmercury borate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- lidocaine gel (Experimental): This group will be those randomized to receiving the intervention with 2% lidocaine gel.
  Interventions: Drug: 2% lidocaine gel
- placebo gel (surgilube) (Placebo Comparator): This group will be randomized to having the intervention with the placebo surgilube gel.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: 2% lidocaine gel — Participants, after informed consent, will be randomized in a 1:1 ratio to the inert gel group or the intervention group. In the intervention group, after tenaculum placement, a Q-tip soaked in approximately 1mL of 2% lidocaine gel will be placed in the cervix up to the level of the internal cervical os. The Q-tip will be held there for 1 minute and then be removed. We will repeat the same procedure in the control group with an inert gel similar in appearance, color and consistency to the lidocaine gel.
  Both the patient and the provider will be blinded to which gel was received. The research assistant will place the gel from its labeled tube into the unlabeled sterile tube in another room.
  Arms: lidocaine gel
Other: placebo — Participants, after informed consent, will be randomized in a 1:1 ratio to the inert gel group or the intervention group. In the intervention group, after tenaculum placement, a Q-tip soaked in approximately 1mL of 2% lidocaine gel will be placed in the cervix up to the level of the internal cervical os. The Q-tip will be held there for 1 minute and then be removed. We will repeat the same procedure in the control/placebo group with an inert gel similar in appearance, color and consistency to the lidocaine gel.
  Both the patient and the provider will be blinded to which gel was received. The research assistant will place the gel from its labeled tube into the unlabeled sterile tube in another room.
  Other Names: surgilube
  Arms: placebo gel (surgilube)

SUMMARY:
The intrauterine device (IUD) is a form of birth control that is extremely effective and safe, even in women who have not yet had children. Women can experience high levels of pain when the IUD is placed inside the uterus, and fear of this pain could be a reason that women decide not to use this method.

This study will randomly (like flipping a coin) assign women who have chosen the IUD as their contraceptive into two groups. One group will have lidocaine anesthetic gel placed into their cervix prior to having the IUD inserted; the other will have an inert gel placed into their cervix instead. The level of pain at three different time points on a 10cm scale and the patient's satisfaction with the procedure will be compared between the two groups to see if using lidocaine gel helps decrease IUD insertional pain

DETAILED DESCRIPTION:
The intrauterine device (IUD) is a highly effective, long-acting, reversible method of contraception used by approximately 8% of women in the developed world. In the United States, historically candidates for IUDs were monogamous, parous women. Recent research has shown that both copper and levonorgestrel IUD use is safe and effective in nulliparous women. Nulliparous and parous women can experience significant amounts of pain during IUD insertion. Concerns about insertional pain could be a barrier to IUD initiation women and their healthcare providers.

This study will recruit women at either the Family Planning Clinic or the offices of Columbia University Family Planning Practice who desire the copper or levonorgestrel IUD for birth control. Women who consent to participating in the study will be randomized to two groups: one group will receive 2% lidocaine gel placed in the cervix prior to IUD placement and the other group will receive a placebo inert gel. The primary objective of this study is to compare the pain scores on a 10cm visual analogue scale in the two groups after tenaculum placement (placing an instrument on the cervix to stabilize it), uterine sounding (measuring of the uterus) and at speculum removal; these are standard procedures during IUD insertion. Secondary outcomes include provider assessment of the patient's pain, patient's level of satisfaction with the insertion, and whether any adverse events such as nausea/vomiting, fainting, or IUD insertion failure occurred.

ELIGIBILITY:
Inclusion Criteria:

* Self-select either a Paragard or Mirena IUD and are appropriate for insertion as determined by their provider
* Age 18-45
* Speak English or Spanish

Exclusion Criteria:

* Lidocaine allergy
* First trimester abortion or miscarriage in the previous six weeks
* Second trimester abortion or miscarriage in the previous 12 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Davis, MD, Principal Investigator — Columbia University
Locations (1):
- Family Planning Clinic / Columbia University Family Planning Practice, New York, New York, United States

REFERENCES:
- [Derived] Maguire K, Davis A, Rosario Tejeda L, Westhoff C. Intracervical lidocaine gel for intrauterine device insertion: a randomized controlled trial. Contraception. 2012 Sep;86(3):214-9. doi: 10.1016/j.contraception.2012.01.005. Epub 2012 Feb 9. PMID 22325115

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine Gel: This group will be those randomized to receiving the intervention with 2% lidocaine gel.
  2% lidocaine gel: Participants, after informed consent, will be randomized in a 1:1 ratio to the inert gel group or the intervention group. In the intervention group, after tenaculum placement, a Q-tip soaked in approximately 1mL of 2% lidocaine gel will be placed in the cervix up to the level of the internal cervical os. The Q-tip will be held there for 1 minute and then be removed. We will repeat the same procedure in the control group with an inert gel similar in appearance, color and consistency to the lidocaine gel.
  Both the patient and the provider will be blinded to which gel was received. The research assistant will place the gel from its labeled tube into the unlabeled sterile tube in another room.
- Placebo Gel (Surgilube): This group will be randomized to having the intervention with the placebo surgilube gel.
  2% lidocaine gel: Participants, after informed consent, will be randomized in a 1:1 ratio to the inert gel group or the intervention group. In the intervention group, after tenaculum placement, a Q-tip soaked in approximately 1mL of 2% lidocaine gel will be placed in the cervix up to the level of the internal cervical os. The Q-tip will be held there for 1 minute and then be removed. We will repeat the same procedure in the control group with an inert gel similar in appearance, color and consistency to the lidocaine gel.
  Both the patient and the provider will be blinded to which gel was received. The research assistant will place the gel from its labeled tube into the unlabeled sterile tube in another room.
Period: Overall Study
Arm/Group | Lidocaine Gel | Placebo Gel (Surgilube)
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Gel | Placebo Gel (Surgilube) | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (6) | 27.6 (6) | 27.4 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 72 | 81 | 153
  Caucasian | 15 | 12 | 27
  Other | 13 | 7 | 20
Parity [Number; unit: participants]
  Nulliparous | 39 | 21 | 60
  Parous | 61 | 79 | 140
Dysmenorrhea [Mean (Standard Deviation); unit: units on a 100mm Visual Analogue Scale] — The 100 mm visual analogue scale measures pain from 0-100. It is a straight line from "no pain" to "worst pain" and it goes from 0 pain on the left to the maximum pain on the right. A higher number reflects more pain. The place where the patient marks her pain is measured from the left and is read as "mm".
  units on a 100mm Visual Analogue Scale | 36.8 (29) | 32.3 (28) | 34.6 (28)
Anticipated pain [Mean (Standard Deviation); unit: units on a 100 mm visual analogue scale] — The 100 mm visual analogue scale measures pain from 0-100. It is a straight line from "no pain" to "worst pain" and it goes from 0 pain on the left to the maximum pain on the right. A higher number reflects more pain. The place where the patient marks her pain is measured from the left and is read as "mm".
  units on a 100 mm visual analogue scale | 56.0 (26) | 57.2 (28) | 56.6 (27)
IUD type [Number; unit: participants]
  Levonogestrel IUD | 30 | 32 | 62
  Copper IUD | 70 | 68 | 138

OUTCOME MEASURES:

1. Primary Outcome: Pain During IUD Insertion at Various Time Points (See Description for Time Points)
Description: Patient marked pain on a 100 mm visual analogue scale during the part of the IUD insertion procedure where the tenaculum was placed, the uterus was measured/sounded, the IUD was inserted into the uterus, and the speculum was removed.
Time Frame: During IUD insertion (see above description for which time points)
Measure: Mean (Standard Deviation); unit: units on a 100 mm visual analogue scale
Arm/Group | Lidocaine Gel | Placebo Gel (Surgilube)
Number analyzed (Participants) | 100 | 100
units on a 100 mm visual analogue scale
  Tenaculum placement | 35.4 (26) | 34.3 (25)
  Uterine sounding | 55.5 (30) | 51.6 (25)
  IUD insertion | 51.0 (31) | 50.9 (32)
  Speculum removal | 20 (43) | 20 (45)

2. Secondary Outcome: Adverse Events
Time Frame: During IUD insertion
Measure: Number; unit: participants
Arm/Group | Lidocaine Gel | Placebo Gel (Surgilube)
Number analyzed (Participants) | 100 | 100
participants
  Nausea | 8 | 4
  Vomiting | 0 | 0
  Dizziness | 9 | 12

3. Secondary Outcome: Provider's Assessment of Patient's Maximum Pain on a Visual Analogue Scale
Description: This secondary analysis looked at provider perception of patient maximum pain during IUD insertion This was not done per intervention because we were looking at the accuracy of the provider's assesment of the patient's pain, which is not dependent on intervention. The provider was blinded to the intervention so that would not have influenced results.
Time Frame: during IUD insertion
Measure: Mean (Standard Deviation); unit: units on a 100 mm visual analogue scale
Groups:
- Participants: The cohort of all 200 women having their IUD inserted.
- Providers: The healthcare provider placing the IUD on that particular participant.
Arm/Group | Participants | Providers
Number analyzed (Participants) | 200 | 200
units on a 100 mm visual analogue scale | 63.8 (27) | 35.3 (26)

ADVERSE EVENTS:
Arm/Group | Lidocaine Gel | Placebo Gel (Surgilube)
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 17/100 | 16/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine Gel (N=100) | Placebo Gel (Surgilube) (N=100)
dizziness (Nervous system disorders) | 9 (9) | 12 (12) — patient was dizzy during the procedure
nausea (Gastrointestinal disorders) | 8 (8) | 4 (4) — patients had some nausea during the procedure (IUD insertion)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes